CLINICAL TRIAL: NCT00789984
Title: Corneal Specular Microscopy in Infectious and Noninfectious Uveitis
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Filipe de Oliveira, UNIFESP
Other Study IDs: CEP1022/07
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Uveitis
Keywords: Keratic precipitates
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: noncontact specular microscopy

SUMMARY:
The purpose of this study is to determine whether some endothelium morphologic variables are different between infectious and noninfectious uveitis group using a noncontact specular microscopy device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infectious and noninfectious uveitis in any activity level and presence of keratic precipitates.

Exclusion Criteria:

* Patients with previous ocular surgery, trauma, contact lens history, corneal dystrophy, corneal edema and high intraocular pressure
* Any other anterior segment disorders affecting the corneal endothelium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infectious and noninfectious uveitis who were attended at local ophthalmology center.
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Oliveira Fd, Oliveira Motta AC, Muccioli C. Corneal specular microscopy in infectious and noninfectious uveitis. Arq Bras Oftalmol. 2009 Jul-Aug;72(4):457-61. doi: 10.1590/s0004-27492009000400006. PMID 19820783